CLINICAL TRIAL: NCT00455221
Title: Safety Assessment of a Peptide Vaccine Derived From Bcr-abl Along With Cytokine Genes in CML Patients Undergoing Imatinib Treatment
Brief Title: Safety Assessment of a Multipeptide-gene Vaccine in CML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 418-A-2209
Record Dates: First submitted 2007-03-31; First posted 2007-04-03 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Leukemia, Myeloid, Chronic
Keywords: CML; Imatinib; vaccine; peptide; gene; MRD; DNA
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peptide Vaccine (Experimental)
  Interventions: Biological: Bcr-abl multipeptide vaccine; Genetic: Cytokine gene adjuvant

INTERVENTIONS:
Biological: Bcr-abl multipeptide vaccine — The first three patients will receive the lower dose of both IL-12 and GM-CSF plasmids. If this is well tolerated, then the next three patients will receive the lower dose of IL-12 plasmid and higher dose of GM-CSF plasmid. If this is well tolerated, then the next three patients will receive the higher dose of IL-12 and lower dose of GM-CSF plasmids. If this is well tolerated, then the next three patients will receive the higher dose of both IL-12 and GM-CSF plasmids. Once assigned to a dose, the patient will receive the same dose throughout their participation in this trial
Genetic: Cytokine gene adjuvant — Cytokine gene adjuvant

SUMMARY:
The primary purpose of this study is to evaluate the safety of a peptide-gene vaccine against CML in patients under Imatinib treatment.

We will also perform some laboratory tests suggesting biological response.

DETAILED DESCRIPTION:
* Patients will continue to take their current dose of Imatinib.
* Patients will undergo HLA-typing to define the HLA A, B, and DR.
* One constant dose of ten bcr-abl peptides (100μg each) will be administered subcutaneously in all patients triweekly for 8 doses.
* Four different doses of IL-12 and GM-CSF plasmids will be tested in this trial. The plasmids will be administered subcutaneously near the vaccination site 24 hours before vaccination.
* The first three patients will receive the lower dose of both IL-12 and GM-CSF plasmids. If this is well tolerated, then the next three patients will receive the lower dose of IL-12 plasmid and higher dose of GM-CSF plasmid. If this is well tolerated, then the next three patients will receive the higher dose of IL-12 and lower dose of GM-CSF plasmids. If this is well tolerated, then the next three patients will receive the higher dose of both IL-12 and GM-CSF plasmids. Once assigned to a dose, the patient will receive the same dose throughout their participation in this trial.
* Each vaccination may consist of one to several shots placed under the skin on the forearm, thigh or trunk area, and the sites will rotate per vaccination.
* During the clinic visit for vaccinations, blood tests will be drawn. If, during the course of therapy, side effects develop that the doctor feels pose a threat to the patient, treatment will be stopped.
* Patients will also undergo DTH skin tests before and after vaccination to see if an immune reaction is occurring at the injection site.
* Patients' lymphocytes will be tested before and after vaccination regarding IFN-γ and IL-4 production to assess immune system activation.
* During the course of treatment we will measure the effect the vaccine is having on the patients CML every three months by:

  1. doing a bone marrow biopsy and aspirate analysis, and
  2. measuring the amount of BCR-ABL that is detectable by RT-PCR in the patients' peripheral blood and bone marrow aspirate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Philadelphia chromosome positive CML who are:

  1. of subtype b3a2
  2. In first complete hematologic response;
  3. have received imatinib for > 12 months of which the last 3 months were at a stable dose of at least 400 mg/day;
  4. have PCR detectable BCR-ABL transcript by qRT-PCR, and
  5. with persistent disease, as defined by <1 log reduction in peripheral blood or bone marrow BCR-ABL transcripts levels compared with a standardized baseline.
* Greater than or equal to 18 years in age
* No known infection with human immunodeficiency virus
* Physician and patient willingness to maintain the baseline dose of imatinib throughout the study period
* Written informed consent obtained from the patient

Exclusion Criteria:

* Female patients who are pregnant or breast feeding or adults of childbearing age who are not using adequate birth control.
* Current use of systemic immunosuppressive medications
* ALT or AST >3X Upper limit Normal
* Prior allogeneic stem cell transplantation
* Other experimental therapy within the past two months
* Prior participation in vaccine studies within the past six months
* Oxygen saturation of less than 95% at room air
* History of recent acute myocardial infarction, unstable angina, or pulmonary decompensation requiring hospitalization within the past 3 months.
* Concurrent and or uncontrolled psychiatric or medical condition which may interfere with the study completion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To assess safety of bcr-abl peptide vaccination in Ph+ or MRD CML patients | At enroll in study and 3 months after intervention

SECONDARY OUTCOMES:
To measure the development of a molecular response to vaccination as measured by 1 log decrease in qRT-PCR BCR-ABL levels for at least 3 months; To measure the development of immune response following vaccination | At enroll in study and 3 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Hamidollah Ghaffari, PhD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Hematology-Oncology & SCT Research Center, Tehran, Tehran Province, Iran